CLINICAL TRIAL: NCT06387966
Title: A Randomized, Double-blind, Placebo-controlled, Dose-escalating, Single-dose, Oral Phase I Clinical Study of the Safety, Tolerability, and Pharmacokinetics of Flonoltinib Maleate Tablets in Healthy Adult Subjects in China
Brief Title: A Phase I Clinical Study of Flonoltinib Maleate Tablets in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Chengdu Zenitar Biomedical Technology Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Other
Other Study IDs: H-FNTN-PI-Ia
Record Dates: First submitted 2024-03-06; First posted 2024-04-29 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Heathly Subjects

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Flonoltinib Maleate Tablets treament group (Experimental): Subjects in this group will take Flonoltinib Maleate Tablets
  Interventions: Drug: Flonoltinib Maleate Tablets
- placebo group (Placebo Comparator): Subjects in this group will take Flonoltinib Maleate Tablets placebo
  Interventions: Drug: Flonoltinib Maleate Tablets placebo

INTERVENTIONS:
Drug: Flonoltinib Maleate Tablets — Day 1 will be used for drug administration, and Day 1~Day 7 will be used for experimental data collection.
  Other Names: 25mg Flonoltinib Maleate Tablets; 50mg Flonoltinib Maleate Tablets; 100mg Flonoltinib Maleate Tablets; 150mg Flonoltinib Maleate Tablets; 200mg Flonoltinib Maleate Tablets
  Arms: Flonoltinib Maleate Tablets treament group
Drug: Flonoltinib Maleate Tablets placebo — Day 1 will be used for drug administration, and Day 1~Day 7 will be used for experimental data collection.
  Other Names: 25mg Flonoltinib Maleate Tablets placebo; 50mg Flonoltinib Maleate Tablets placebo; 100mg Flonoltinib Maleate Tablets placebo; 150mg Flonoltinib Maleate Tablets placebo; 200mg Flonoltinib Maleate Tablets placebo
  Arms: placebo group

SUMMARY:
Evaluate the safety , tolerability and pharmacokinetics of Flonoltinib Maleate tablets in a single increasing dose oral administered to healthy adult Chinese subjects.Subjects will divide into experimental group and placebo group, conduct single oral administration safety and tolerability test group by group.

ELIGIBILITY:
Inclusion Criteria:

1. Age and gender: 18 to 45 years old (including 18 and 45 years old), no gender limit;
2. The weight of male subjects is ≥50.0 kg, the weight of female subjects is ≥45.0 kg, and the body mass index (BMI) is between 19.0 and 25.0 kg/m2 (including the boundary value);
3. Those who fully understand the trial content, trial drugs, trial process, etc., can communicate well with the researchers, are willing to comply with the research regulations, voluntarily participate in the trial and sign the informed consent form.

Exclusion Criteria:

1. Those with a history of severe allergies (such as angioedema and anaphylactic shock), allergies (such as allergies to pollen, two or more drugs/foods), or those with Those who are judged by the researcher to have a clinically significant history of food or drug allergies or other allergic diseases (asthma, urticaria, eczematous dermatitis, etc.); or those who are known to be allergic to JAK inhibitors or to excipients contained in the trial drug ;
2. Pre-selection physical examination, vital signs, 12-lead electrocardiogram, laboratory tests (including: blood routine, blood biochemistry, urine routine, blood pregnancy (females only), infectious disease screening, antinuclear antibodies, coagulation function , tuberculosis antibodies, chest anteroposterior X-ray examination, abdominal color ultrasound) results are abnormal and clinically significant;
3. QTcF > 440 ms for males and > 460 ms for females on ECG during the screening period;
4. Those who have undergone major surgical operations within 3 months before screening or plan to undergo surgery during the trial;
5. Those who suffer from acute diseases within 2 weeks before screening; those who have clinically significant infections (such as upper respiratory tract infection, nasopharyngitis, urinary system infection, etc.) within 3 months before screening; those who have any symptoms within 7 days before screening Those with evidence of infection; those with a history of herpes simplex infection or recurrent (>1) herpes zoster or disseminated herpes zoster.
6. Have any history of serious clinical diseases or diseases or conditions that the researcher believes may affect the test results, including but not limited to the circulatory system, endocrine system, nervous system, digestive system, urinary system or History of blood, immune, psychiatric and metabolic diseases;
7. Those with a history of dysphagia or any gastrointestinal system disease (or gastrointestinal resection, etc.) that affects drug absorption;
8. Those with irregular bowel movements and habitual constipation or diarrhea;
9. Those with a history of lipid metabolism defects, such as: familial hyperlipidemia, lipoid nephropathy, or patients with acute pancreatitis accompanied by hyperlipidemia, etc.;
10. Those whose urine is positive for multiple combined drug tests (including morphine, methamphetamine, ketamine, methylenedioxyamphetamine, and tetrahydrocannabinolic acid);
11. Those who have a history of drug abuse or drug dependence;
12. Those who have been vaccinated within 8 weeks before screening, or plan to be vaccinated during the study or within 8 weeks after the administration of study drugs;
13. Those who have donated blood or lost ≥400 mL of blood or received blood transfusions within 3 months before screening; or those who have donated blood or blood components within 1 month after the planned trial ends;
14. Those who have special requirements for diet or cannot comply with the unified diet and corresponding regulations of the research center;
15. Those who smoke more than 3 cigarettes/day or the same amount of tobacco within 3 months before screening; or drink ≥14 units of alcohol per week (1 unit is equal to 17.5mL or 14g of pure alcohol, Approximately equal to 35mL of 50° liquor or 350mL of 5° beer); or those who do not agree to abstain from smoking or drinking during the trial; or those whose alcohol breath test results are positive;
16. Those who have taken any prescription drugs, over-the-counter drugs, any vitamin products or Chinese herbal medicines (JAK inhibitors, immunosuppressants, etc.) within 14 days before screening;
17. Concomitant use of strong inducers of liver metabolic enzymes (such as: omeprazole, barbiturates, carbamazepine, aminolutamide) within 4 weeks (28 days) before screening (e.g., griseofulvin, methamphetamine, phenytoin, glutamidate, rifampicin, sulfinpyrazone, roxithromycin, etc.), or others judged by the investigator to be likely to affect the pharmacokinetics of the test drug in vivo Medication history learner. Those who have taken any drugs known to cause QT/QTcF interval prolongation or drugs with a risk of causing torsade de pointes (TdP) within 4 weeks (28 days) before screening; or those with long half-life;
18. Within 48 hours before administration, consumption of any food or beverage containing caffeine (such as coffee, strong tea, cola, chocolate, etc.), or containing grapefruit juice, etc. may affect metabolism. Foods that may affect enzymes, or those who consume alcoholic foods or drinks;
19. Those who participated in other clinical trials and used investigational drugs, vaccines or devices within 3 months before the first dose;
20. Pregnant or lactating women or women of childbearing age who have had unprotected sexual intercourse within 14 days before screening;
21. During the trial, the subject or his partner is unwilling to use non-drug contraceptive methods (such as complete abstinence, condoms, IUDs, sterilization, etc.) for contraception or after administration of study drugs The subject and/or his or her partner have pregnancy plans within 3 months;
22. The subject may not be able to complete the study due to other reasons or the researcher may think there are other factors that make him or her unsuitable to participate in the trial.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2024-03-18 (Actual); Primary Completion 2024-08-15 (Actual); Study Completion 2024-08-15 (Actual)

PRIMARY OUTCOMES:
Tmax | Day1 Within 30 minutes before administration and 15 minutes, 0.5 hours, 1 hours, 2 hours, 2.5 hours, 3 hours, 3.5 hours, 4 hours, 5hours, 6 hours, 8 hours, 12 hours, 24 hours, 48 hours, 72 hours, 96 hours, 120 hours, 144 hours after administration
  time to peak
Cmax | Day1 Within 30 minutes before administration and 15 minutes, 0.5 hours, 1 hours, 2 hours, 2.5 hours, 3 hours, 3.5 hours, 4 hours, 5hours, 6 hours, 8 hours, 12 hours, 24 hours, 48 hours, 72 hours, 96 hours, 120 hours, 144 hours after administration
  maximum concentration
t1/2 | Day1 Within 30 minutes before administration and 15 minutes, 0.5 hours, 1 hours, 2 hours, 2.5 hours, 3 hours, 3.5 hours, 4 hours, 5hours, 6 hours, 8 hours, 12 hours, 24 hours, 48 hours, 72 hours, 96 hours, 120 hours, 144 hours after administration
  Terminal phase elimination half-life
CL/F | Day1 Within 30 minutes before administration and 15 minutes, 0.5 hours, 1 hours, 2 hours, 2.5 hours, 3 hours, 3.5 hours, 4 hours, 5hours, 6 hours, 8 hours, 12 hours, 24 hours, 48 hours, 72 hours, 96 hours, 120 hours, 144 hours after administration
  Apparent clearance rate
AUC0-t | Day1 Within 30 minutes before administration and 15 minutes, 0.5 hours, 1 hours, 2 hours, 2.5 hours, 3 hours, 3.5 hours, 4 hours, 5hours, 6 hours, 8 hours, 12 hours, 24 hours, 48 hours, 72 hours, 96 hours, 120 hours, 144 hours after administration
  Area under the blood concentration-time curve from 0 o 'clock to the last measurable concentration at collection time t
AUC0-∞ | Day1 Within 30 minutes before administration and 15 minutes, 0.5 hours, 1 hours, 2 hours, 2.5 hours, 3 hours, 3.5 hours, 4 hours, 5hours, 6 hours, 8 hours, 12 hours, 24 hours, 48 hours, 72 hours, 96 hours, 120 hours, 144 hours after administration
  The area under the blood drug concentration-time curve from 0 to infinity time
Vz/F | Day1 Within 30 minutes before administration and 15 minutes, 0.5 hours, 1 hours, 2 hours, 2.5 hours, 3 hours, 3.5 hours, 4 hours, 5hours, 6 hours, 8 hours, 12 hours, 24 hours, 48 hours, 72 hours, 96 hours, 120 hours, 144 hours after administration
  apparent volume of distribution
Ae0-144hours and Ae% | Day1 Within 2hours before administration and 0~4 hours, 4~8 hours, 8~12 hours, 12~24 hours, 24~36 hours, 36~48 hours, 48~72 hours, 72~96hours, 96~120 hours, 120~144 hours after administration
  The pharmacokinetic statistical parameters of urine are the cumulative excretion (Ae0-144hours) and excretion rate (Ae%) of prototype drugs and major metabolites in urine，that is collected from the 50 mg and 150mg dose groups.
Ae0-144hours and Ae% | 1 blank fecal sample before administration and after administration: 0~24 hours, 24~48 hours,48~72 hours, 72~96hours, 96~120 hours, 120~144 h ours
  The statistical parameters of fecal pharmacokinetics are the cumulative excretion of prototype drugs and major metabolites in feces (Ae0-144hours) and excretion rate (Ae%) ,that is collected from the 50 mg and 150mg dose groups

SECONDARY OUTCOMES:
security indicators | According to the experimental schedule D-14-D7 or early termination
  Observe the changes in vital signs, physical examination, clinical symptoms, laboratory tests, ECG, and occurrence of adverse events of the subjects after medication.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaolan Yong, bachelor, Principal Investigator — Chengdu Xinhua Hospital
Locations (1):
- Chengdu Xinhua Hospital, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No